CLINICAL TRIAL: NCT05072756
Title: Opinion of Brazilian Gynecologists on Hormone Therapy for Menopause and Prescriptive
Brief Title: Opinion of Brazilian Gynecologists on Hormone Therapy for Menopause and Prescriptive Habits
Status: Completed | Type: Observational
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Luciano de Melo Pompei', Auxiliary Professor at Gynecology Department, Faculdade de Medicina do ABC
Other Study IDs: 40147120.8.0000.0082
Record Dates: First submitted 2021-09-17; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Menopause; Opinions; Hormone Replacement Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gynecologists: Brazilian gynecologists who agreed to participate and answered the questionnaire
  Interventions: Other: Applying a questionnaire

INTERVENTIONS:
Other: Applying a questionnaire — The participants have to answer a questionnaire addressing their opinion on menopausal hormone replacement therapy

SUMMARY:
To evaluate Brazilian gynecologists, through structured online questionnaires, with questions directed to their opinions and prescriptive habits about menopause hormone therapy. Research participants will complete the questionnaires in digital format online.

DETAILED DESCRIPTION:
There are few Brazilian population studies on the opinion of Brazilian gynecologists about the hormonal therapy of menopause in climacteric women, their prescriptive habits and their views on the availability of treatments offered, demanding better evaluation and justifying efforts to analyze the perception of professionals in this area in our country.

Methods: To assess gynecologists across the country, through structured online questionnaires, with questions aimed at knowing their opinions and prescriptive habits about menopause hormone therapy. Research participants will complete the questionnaires in digital format online. Doctors will be invited to participate by e-mail messages and by social media.

ELIGIBILITY:
Inclusion Criteria:

* Brazilian licensed gynecologist doctors

Exclusion Criteria:

* Retired doctors
* Health professionals other than medicine doctor
* Medical specialties other than Gynecology
* Medical employees of the pharmaceutical industry

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Active Brazilian licensed gynecologist doctors who see patients
Sampling Method: Non-Probability Sample
Enrollment: 1339 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2021-09-04 (Actual)

PRIMARY OUTCOMES:
Prescription preference | At Day 1
  Answer to the questionnaire addressing gynecologists' prescription habit for menopausal women

SECONDARY OUTCOMES:
Knowledge of window of opportunity for hormone replacement therapy | At Day 1
  This is to see which proportion of gynecologists know the principle of window of opportunity for menopausal hormone replacement therapy
Knowledge of indications and contraindications of hormone replacement therapy | At Day 1
  This is to see which proportion of gynecologists know the indications and contraindicationsv of menopausal hormone replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Luciano M Pompei, Principal Investigator — Faculdade de Medicina do ABC
Locations (1):
- Centro de Atenção Integral à Saúde da Mulher, São Bernardo do Campo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
This is not an interventional study, so, the researches understand that there is no reason to share individual participant data.

REFERENCES:
- [Background] Taylor HS, Kagan R, Altomare CJ, Cort S, Bushmakin AG, Abraham L. Knowledge of clinical trials regarding hormone therapy and likelihood of prescribing hormone therapy. Menopause. 2017 Jan;24(1):27-34. doi: 10.1097/GME.0000000000000711. PMID 27575548
- [Background] Buhling KJ, von Studnitz FS, Jantke A, Eulenburg C, Mueck AO. Use of hormone therapy by female gynecologists and female partners of male gynecologists in Germany 8 years after the Women's Health Initiative study: results of a survey. Menopause. 2012 Oct;19(10):1088-91. doi: 10.1097/gme.0b013e318250bfda. PMID 22692331
- [Background] Yeganeh L, Boyle J, Teede H, Vincent A. Knowledge and attitudes of health professionals regarding menopausal hormone therapies. Climacteric. 2017 Aug;20(4):348-355. doi: 10.1080/13697137.2017.1304906. Epub 2017 Apr 5. PMID 28379046